CLINICAL TRIAL: NCT01152515
Title: A Low Dose Remifentanil Infusion During Tracheal Extubation in Surgical Intensive Care Unit Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, MD, PhD, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 4-2010-0022
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Tracheal Extubation
Keywords: safety and efficacy of maintaining a remifentanil infusion during extubation in propofol-remifentanil sedated patients after surgery
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (No Intervention): stopping of propofol and remifentanil infusion
- Remifentanil (Active Comparator): stopping of propofol and maintenance of remifentanil infusion
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Control group : stopping of propofol and remifentanil infusion Remifentanil group : stopping of propofol and maintenance of remifentanil infusion
  Arms: Remifentanil

SUMMARY:
Tracheal extubation can be associated with hyperdynamic circulatory response. The investigators examined the effect of maintaining a remifentanil infusion on the cardiovascular response during extubation in propofol-remifentanil sedated patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20
2. Short term ventilator care after surgery in intensive care unit

Exclusion Criteria:

1. pneumonia
2. chronic obstructive lung disease
3. asthma
4. end stage renal disease
5. risk factors for aspiration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Remifentanil
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Remifentanil | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 58 (13) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure Changes During Extubation
Time Frame: 10 min
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Remifentanil
Number analyzed (Participants) | 25 | 25
mmHg
  5 min after extuabtion | 94 (17) | 97 (13)
  10 min after extubation | 96 (17) | 97 (13)

2. Secondary Outcome: Time of Awake
Description: Time of BIS > 80 : time between 'stopping of propofol'
Time Frame: 1 hour
Measure: Median (Full Range); unit: min
Arm/Group | Control | Remifentanil
Number analyzed (Participants) | 25 | 25
min | 3.5 [1 to 10] | 4 [1 to 10]

3. Primary Outcome: HR Changes During Extubation
Time Frame: 10 min
Measure: Mean (Standard Deviation); unit: beat/min
Arm/Group | Control | Remifentanil
Number analyzed (Participants) | 25 | 25
beat/min
  5 min after extubation | 94 (18) | 95 (13)
  10 min after extubation | 94 (17) | 93 (12)

4. Primary Outcome: The Grade of Coughing During Extubation
Description: Grade of cough was assessed on a four-point scale (0=no coughing, 1=single cough, 2=more than one episode of nonsustained coughing, 3=sustained and repetitive coughing with head lift).
Time Frame: 2 min
Measure: Number; unit: participants
Arm/Group | Control | Remifentanil
Number analyzed (Participants) | 25 | 25
participants
  0 | 8 | 11
  1 | 11 | 9
  2 | 4 | 3
  3 | 2 | 2

5. Secondary Outcome: Time of Extubation
Description: Time of extubation : time between 'stopping of propofol' and 'extubation'
Time Frame: 1 hr
Measure: Median (Full Range); unit: min
Arm/Group | Control | Remifentanil
Number analyzed (Participants) | 25 | 25
min | 8 [4 to 17] | 14 [3 to 40]

ADVERSE EVENTS:
Arm/Group | Control | Remifentanil
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No